CLINICAL TRIAL: NCT02533115
Title: Expanded Access Protocol of CPX-351 (Cytarabine:Daunorubicin) Liposome Injection for Patients 60-75 Years of Age With Secondary AML
Brief Title: EAP of CPX-351 (VYXEOS) for Patients 60-75 Years of Age With Secondary AML
Acronym: 401
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CLTR0314-401
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Secondary AML
Keywords: VYXEOS
MeSH Terms: interventions — CPX-351

INTERVENTIONS:
Drug: CPX-351 — CPX-351 (cytarabine:daunorubicin) Liposome for Injection is a liposomal formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin. The two drugs are present inside the liposome in a 5:1 molar ratio shown to act synergistically in pre-clinical studies. The liposome membrane is composed of distearoylphosphatidylcholine, distearoylphosphatidylglycerol and cholesterol in a 7:2:1 molar ratio.
  CPX-351 is provided as a sterile, pyrogen-free, purple, lyophilized product in 50 mL glass, single-use vials. Each 50 mL vial after reconstitution contains 20 mL of CPX-351 (5 units/mL). Each unit (u) contains 1 mg cytarabine and 0.44 mg daunorubicin base in liposomes suspended in sucrose. Product is stored at 5˚ ± 3PoPC.

SUMMARY:
This study is a Phase IV Expanded Access Protocol (EAP) of CPX-351 in patients with secondary acute myeloid leukemia who are suitable for treatment with intensive chemotherapy.

DETAILED DESCRIPTION:
The hypothesis that CPX-351 treatment may be safe and efficacious in patients with newly diagnosed secondary AML comes from a single randomized Phase II study which observed significant improvement in survival in a 52-patient subset of patients with secondary AML. A Phase III confirmatory study has recently completed accrual and final results are not expected until mid-2016. Therefore, the sponsor has chosen to make CPX-351 available to secondary AML patients through this expanded access protocol until commercialization of CPX-351 or more information about the clinical utility is known.

This study is a Phase IV multicenter, single-arm open-label Expanded Access Protocol (EAP) of CPX-351 in patients with secondary acute myeloid leukemia who are suitable for treatment with intensive chemotherapy. Patients may receive up to two inductions and four consolidation courses. Patients will be monitored for safety (early deaths, serious adverse events, grade 3 and 4 adverse events, etc.) while on the study and for SAEs for 30 days after the last dose of CPX-351. Study enrollment will be available through commercialization of CPX-351.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily give informed consent
* Age 60- 75 years
* Pathological diagnosis of AML according to WHO criteria (with at least 20% blasts in the peripheral blood or bone marrow)
* Confirmation of:

  * Therapy related AML: t-AML must have a history of prior cytotoxic therapy or ionizing radiotherapy for an unrelated disease
  * AML with a history of myelodysplasia
  * AML with a history of CMMoL
  * De novo AML with karyotypic abnormalities characteristic of MDS per WHO (see table)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Laboratory values fulfilling the following:

  * Serum creatinine < 2.0 mg/dL
  * Serum total bilirubin < 2.0 mg/dL
  * Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN Note: If elevated liver enzymes above the ULN are related to disease, higher levels of ALT and AST may be considered.
* Cardiac ejection fraction ≥ 50% by echocardiography or MUGA

Exclusion Criteria:

* Except for CMMoL, patients with history of myeloproliferative neoplasms (MPN) (defined as a history of essential thrombocytosis or polycythemia vera, or idiopathic myelofibrosis prior to the diagnosis of AML) or combined MDS/MPN are not eligible.
* Acute promyelocytic leukemia [t(15;17)] or favorable cytogenetics, including t(8;21) or inv16 if known at the time of registration.
* Clinical evidence of active CNS leukemia
* Patients with active (uncontrolled, metastatic) second malignancies are excluded.
* In the event of rapidly proliferative disease use of hydroxyurea is permitted until 24 hours before the start of study treatment.
* Any major surgery or radiation therapy within four weeks.
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/mP2P daunorubicin (or equivalent).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Patients with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
* Active or uncontrolled infection. Patients with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs.
* Current evidence of invasive fungal infection (blood or tissue culture); patients with recent fungal infection must have post treatment negative culture(s) to be eligible; known HIV (new testing not required) or evidence of active hepatitis B or C infection (with rising transaminase values)
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-metabolism disorder

Ages: 60 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Northside Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - The University of Kansas Hospital, Kansas City, Kansas
  - Weill Cornell Medical College- NY Presbyterian Hospital, New York, New York

REFERENCES:
- [Derived] Roboz GJ, Larson ML, Rubenstein SE, Solomon SR, Schiller GJ, An Q, Chiarella M, Louie AC, Lin TL. Final safety and efficacy results from the CPX-351 early access program for older patients with high-risk or secondary acute myeloid leukemia. Leuk Lymphoma. 2020 May;61(5):1188-1194. doi: 10.1080/10428194.2020.1725503. Epub 2020 Feb 26. PMID 32102577